CLINICAL TRIAL: NCT00820027
Title: A Phase III Randomized, Double-Blind, Placebo- and Active-Comparator-Controlled, Multiple-Dose, Clinical Trial to Study the Safety and Efficacy of MK0663/Etoricoxib and Ibuprofen in the Treatment of Postorthopedic Knee Replacement Surgery Pain
Brief Title: Study of MK-0663/Etoricoxib in Postorthopedic Knee Replacement Surgery Pain (MK-0663-098)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Organon and Co (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 0663-098; 2009_502 (Other: Merck Registration Number)
Record Dates: First submitted 2009-01-07; First posted 2009-01-09 (Estimated); Results first posted 2020-04-07 (Actual); Last update posted 2022-02-09 (Actual); Status verified 2022-02

CONDITIONS: Pain, Postoperative
MeSH Terms: conditions — Pain, Postoperative | interventions — Etoricoxib; Ibuprofen; Morphine; Oxycodone

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- Etoricoxib 90 mg (Experimental): Participants received etoricoxib 90 mg once daily, matching placebo to etoricoxib 120 mg once daily, and matching placebo to ibuprofen 600 mg every 8 hours for 7 days.
  Interventions: Drug: Etoricoxib 90 mg; Drug: Matching Placebo for Etoricoxib 120 mg; Drug: Matching Placebo for Ibuprofen; Drug: Morphine; Drug: Oxycodone
- Etoricoxib 120 mg (Experimental): Participants received etoricoxib 120 mg once daily, matching placebo to etoricoxib 90 mg once daily, and matching placebo to ibuprofen 600 mg every 8 hours for 7 days.
  Interventions: Drug: Etoricoxib 120 mg; Drug: Matching Placebo for Etoricoxib 90 mg; Drug: Matching Placebo for Ibuprofen; Drug: Morphine; Drug: Oxycodone
- Ibuprofen 1800 mg (Active Comparator): Participants received ibuprofen 600 mg every 8 hours, matching placebo to etoricoxib 120 mg once daily, and matching placebo to etoricoxib 90 mg once daily for 7 days.
  Interventions: Drug: Ibuprofen 600 mg; Drug: Matching Placebo for Etoricoxib 120 mg; Drug: Matching Placebo for Etoricoxib 90 mg; Drug: Morphine; Drug: Oxycodone
- Placebo (Placebo Comparator): Participants received matching placebo to etoricoxib 90 mg and matching placebo to etoricoxib 120 mg once daily, and matching placebo to ibuprofen every 8 hours for 7 days.
  Interventions: Drug: Matching Placebo for Etoricoxib 120 mg; Drug: Matching Placebo for Etoricoxib 90 mg; Drug: Matching Placebo for Ibuprofen; Drug: Morphine; Drug: Oxycodone

INTERVENTIONS:
Drug: Etoricoxib 90 mg — One 90 mg tablet once daily
  Other Names: MK-0663
  Arms: Etoricoxib 90 mg
Drug: Etoricoxib 120 mg — Two 60 mg tablets once daily
  Other Names: MK-0663
  Arms: Etoricoxib 120 mg
Drug: Ibuprofen 600 mg — One tablet three times daily
  Arms: Ibuprofen 1800 mg
Drug: Matching Placebo for Etoricoxib 120 mg — Two tablets once daily
  Arms: Etoricoxib 90 mg; Ibuprofen 1800 mg; Placebo
Drug: Matching Placebo for Etoricoxib 90 mg — One tablet once daily
  Arms: Etoricoxib 120 mg; Ibuprofen 1800 mg; Placebo
Drug: Matching Placebo for Ibuprofen — One tablet three times daily
  Arms: Etoricoxib 120 mg; Etoricoxib 90 mg; Placebo
Drug: Morphine — As needed via patient-controlled analgesia (PCA) device or as a bolus intravenous injection
Drug: Oxycodone — 5 mg as needed

SUMMARY:
The purpose of this study was to evaluate the efficacy and safety of Etoricoxib compared to placebo and ibuprofen in the treatment of postoperative pain associated with unilateral total knee replacement surgery. The hypotheses for this study were that the average pain intensity difference (at rest) in participants treated with Etoricoxib (120 mg, 90 mg) is superior to placebo, the average total daily dose of morphine in participants treated with Etoricoxib (120 mg, 90 mg) is less than in participants treated with placebo, and that Etoricoxib (120 mg, 90 mg) will be generally safe and well tolerated by participants treated for pain following total knee replacement orthopedic surgery.

ELIGIBILITY:
Inclusion Criteria:

- Is in generally good health and is scheduled to have a total knee replacement

Exclusion Criteria:

* Is allergic, intolerant to, or has a history of a significant clinical or laboratory adverse experience associated with etoricoxib or other cyclooxygenase-2 (COX-2) inhibitors/non-steroidal anti-inflammatory drugs (NSAIDs), ibuprofen, morphine, or oxycodone, or has hypersensitivity to aspirin, or other NSAIDs
* Has uncontrolled hypertension
* Is currently a user of any illicit drugs, or has a history of drug or alcohol abuse within the past 5 years

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 776 (Actual)
Dates: Start 2008-12-15 (Actual); Primary Completion 2010-12-13 (Actual); Study Completion 2010-12-14 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC

REFERENCES:
- [Derived] Rawal N, Viscusi E, Peloso PM, Minkowitz HS, Chen L, Shah S, Mehta A, Chitkara DK, Curtis SP, Papanicolaou DA. Evaluation of etoricoxib in patients undergoing total knee replacement surgery in a double-blind, randomized controlled trial. BMC Musculoskelet Disord. 2013 Oct 24;14:300. doi: 10.1186/1471-2474-14-300. PMID 24156640

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Etoricoxib 90 mg | Etoricoxib 120 mg | Ibuprofen 1800 mg | Placebo
Started | 224 | 230 | 224 | 98
Completed | 198 | 216 | 203 | 85
Not Completed | 26 | 14 | 21 | 13
Not completed — Adverse Event | 15 | 8 | 10 | 5
Not completed — Lack of Efficacy | 2 | 1 | 2 | 2
Not completed — Physician Decision | 0 | 1 | 1 | 0
Not completed — Protocol Violation | 3 | 0 | 4 | 0
Not completed — Withdrawal by Subject | 6 | 4 | 4 | 6

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Etoricoxib 90 mg | Etoricoxib 120 mg | Ibuprofen 1800 mg | Placebo | Total
Number analyzed (Participants) | 224 | 230 | 224 | 98 | 776
Age, Continuous [Mean (Standard Deviation); unit: years] | 65.7 (8.5) | 64.7 (8.1) | 66.0 (8.1) | 65.2 (7.9) | 65.4 (8.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 134 | 139 | 152 | 56 | 481
  Male | 90 | 91 | 72 | 42 | 295
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 6 | 1 | 2 | 1 | 10
  Not Hispanic or Latino | 218 | 229 | 222 | 97 | 766
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 1 | 0 | 1
  Asian | 22 | 14 | 20 | 4 | 60
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 8 | 2 | 2 | 2 | 14
  White | 190 | 212 | 199 | 92 | 693
  More than one race | 3 | 1 | 2 | 0 | 6
  Unknown or Not Reported | 1 | 1 | 0 | 0 | 2

OUTCOME MEASURES:

1. Primary Outcome: Average Change From Baseline for Pain Intensity at Rest Over Days 1 to 3 (Etoricoxib vs. Placebo)
Description: The pain intensity difference was measured at rest over Days 1 through 3 in patients treated with etoricoxib (120 mg, 90 mg) compared to placebo for the treatment of pain following total knee replacement orthopedic surgery. Pain intensity difference at rest was measured on a numerical rating scale (NRS) from 0 - 10 points (0=no pain, to 10=pain as bad as you can imagine). Comparison to placebo was conducted in a step-down manner (the 90-mg dose was evaluated only if the null hypotheses for co-primary endpoints [Pain Intensity Difference (PID) and Morphine] 120-mg doses were rejected). The primary analyses for change from baseline in average pain intensity at rest over Days 1 to 3 was performed using the longitudinal data analysis (LDA) method with the terms for baseline pain intensity (moderate or severe), type of anesthesia (spinal or general), treatment, day, and the interaction of day by treatment.
Time Frame: Baseline and Days 1-3
Population: All randomized participants, excluding those who didn't receive at least 1 dose of study treatment, lacked 1 post-randomization measurement, were randomized at a specific site, or received continuous infusion of morphine by patient control analgesia (PCA). Per protocol, the ibuprofen arm was not included in this outcome measure.
Measure: Least Squares Mean (95% Confidence Interval); unit: Score on a scale
Arm/Group | Etoricoxib 90 mg | Etoricoxib 120 mg | Placebo
Number analyzed (Participants) | 211 | 224 | 96
Score on a scale | -3.93 [-4.17 to -3.69] | -3.87 [-4.11 to -3.64] | -3.39 [-3.74 to -3.04]
Statistical Analysis 1: Comparison: Etoricoxib 120 mg vs Placebo; Test type: Superiority; p = 0.018, longitudinal data analysis (LDA); Estimate from LDA model with terms for baseline pain intensity, type of anesthesia, treatment, day, and interaction of day by treatment; Difference in Least Squares Mean = -0.49, 95% CI 2-sided [-0.89 to -0.08]
Statistical Analysis 2: Comparison: Etoricoxib 90 mg vs Placebo; Test type: Superiority; p = 0.009, LDA; [statistical method as in outcome 1, analysis 1]; Difference in Least Squares Mean = -0.54, 95% CI 2-sided [-0.95 to -0.14]

2. Primary Outcome: Average Total Daily Dose of Postoperative Morphine Over Days 1 to 3 (Etoricoxib vs. Placebo)
Description: The average total dose of morphine was assessed when participant received etoricoxib 120 milligram(mg)/90 mg compared to placebo. Opioids taken were converted to mg morphine equivalents according to the following conventions: 1 mg morphine sulphate=1 mg morphine,1 mg morphine hydrochloride=1.17 mg morphine. A 5 mg oxycodone tablet=2.5 mg morphine,12.5 mg meperidine =1.67 mg morphine. Least-squares mean back-transformed; estimate obtained from longitudinal analysis of variance (ANOVA) model on log-transformed morphine dose with terms for baseline pain intensity(moderate or severe),type of anesthesia (spinal, general), treatment, day, and the interaction of day by treatment.
Time Frame: Days 1-3
Population: All randomized participants, excluding those who didn't receive at least 1 dose of study treatment, lacked 1 post-randomization measurement, were randomized at a specific site, or received continuous infusion of morphine by PCA. Per protocol, the ibuprofen arm was not included in this outcome measure.
Measure: Geometric Least Squares Mean (95% Confidence Interval); unit: milligrams (mg)
Arm/Group | Etoricoxib 90 mg | Etoricoxib 120 mg | Placebo
Number analyzed (Participants) | 215 | 225 | 96
milligrams (mg) | 8.87 [7.88 to 9.97] | 9.25 [8.26 to 10.40] | 13.40 [11.20 to 16.00]
Statistical Analysis 1: Comparison: Etoricoxib 120 mg vs Placebo; Test type: Superiority; p < 0.001, ANOVA; Estimate from ANOVA model with terms for baseline pain intensity, type of anesthesia, treatment, day, and interaction of day by treatment; Between-Treatment Ratio = 0.69, 95% CI 2-sided [0.56 to 0.85] — A ratio <1 indicates a beneficial effect of Etoricoxib
Statistical Analysis 2: Comparison: Etoricoxib 90 mg vs Placebo; Test type: Superiority; p < 0.001, ANOVA; [statistical method as in outcome 2, analysis 1]; Between-Treatment Ratio = 0.66, 95% CI 2-sided [0.54 to 0.82] — A ratio <1 indicates a beneficial effect of Etoricoxib

3. Primary Outcome: Percentage of Participants With at Least One Adverse Event of Congestive Heart Failure, Pulmonary Edema, or Cardiac Failure
Description: An adverse event (AE) is defined as any unfavorable and unintended change in the structure, function, or chemistry of the body temporally associated with the use of the study product, whether or not considered related to the use of the product. Any worsening (i.e., any clinically significant adverse change in frequency and/or intensity) of a preexisting condition which is temporally associated with the use of the study product, is also an AE.
Time Frame: Up to 21 days
Population: The analysis population consisted of all randomized patients who received at least one dose of study treatment.
Measure: Number; unit: Percentage of Participants
Arm/Group | Etoricoxib 90 mg | Etoricoxib 120 mg | Ibuprofen 1800 mg | Placebo
Number analyzed (Participants) | 222 | 230 | 223 | 98
Percentage of Participants | 0.5 | 0.0 | 0.0 | 0.0
Statistical Analysis 1: Comparison: Etoricoxib 90 mg vs Placebo; Test type: Other; p = 0.506, Miettinen & Nurminen; Difference in Percent = 0.5, 95% CI 2-sided [-3.3 to 2.5]
Statistical Analysis 2: Comparison: Etoricoxib 120 mg vs Placebo; Test type: Other; p > 0.999, Miettinen & Nurminen; Difference in Percent = 0.0, 95% CI 2-sided [-3.8 to 1.7]
Statistical Analysis 3: Comparison: Ibuprofen 1800 mg vs Placebo; Test type: Other; p > 0.999, Miettinen & Nurminen; Difference in Percent = 0.0, 95% CI 2-sided [-3.8 to 1.7]
Statistical Analysis 4: Comparison: Etoricoxib 90 mg vs Ibuprofen 1800 mg; Test type: Other; p = 0.316, Miettinen & Nurminen; Difference in Percent = 0.5, 95% CI 2-sided [-1.3 to 2.5]
Statistical Analysis 5: Comparison: Etoricoxib 120 mg vs Ibuprofen 1800 mg; Test type: Superiority; p > 0.999, Miettinen & Nurminen; Difference in Percent = 0.0, 95% CI 2-sided [-1.7 to 1.7]
Statistical Analysis 6: Comparison: Placebo; Placebo vs. Ibuprofen 1800 mg; Test type: Other; p > 0.999, Miettinen & Nurminen; Difference in Percent = 0.0, 95% CI 2-sided [-1.7 to 3.8]
Statistical Analysis 7: Comparison: Etoricoxib 90 mg vs Etoricoxib 120 mg; Test type: Other; p = 0.309, Miettinen & Nurminen; Difference in Percent = -0.5, 95% CI 2-sided [-2.5 to 1.2]

4. Primary Outcome: Percentage of Participants With at Least One Edema-Related AE
Description: An AE is defined as any unfavorable and unintended change in the structure, function, or chemistry of the body temporally associated with the use of the study product, whether or not considered related to the use of the product. Any worsening (i.e., any clinically significant adverse change in frequency and/or intensity) of a preexisting condition which is temporally associated with the use of the study product, is also an AE. Edema is swelling caused by excess fluid trapped in body tissues.
Time Frame: Up to 21 days
Population: The analysis population consisted of all randomized patients who received at least one dose of study treatment.
Measure: Number; unit: Percentage of Participants
Arm/Group | Etoricoxib 90 mg | Etoricoxib 120 mg | Ibuprofen 1800 mg | Placebo
Number analyzed (Participants) | 222 | 230 | 223 | 98
Percentage of Participants | 0.9 | 1.7 | 1.8 | 4.1
Statistical Analysis 1: Comparison: Etoricoxib 90 mg vs Placebo; Test type: Other; p = 0.054, Miettinen & Nurminen; Difference in Percent = -3.2, 95% CI 2-sided [-9.2 to 0.1]
Statistical Analysis 2: Comparison: Etoricoxib 120 mg vs Placebo; Test type: Other; p = 0.209, Miettinen & Nurminen; Difference in Percent = -2.3, 95% CI 2-sided [-8.4 to 1.2]
Statistical Analysis 3: Comparison: Ibuprofen 1800 mg vs Placebo; Test type: Other; p = 0.227, Miettinen & Nurminen; Difference in Percent = -2.3, 95% CI 2-sided [-8.4 to 1.3]
Statistical Analysis 4: Comparison: Etoricoxib 90 mg vs Ibuprofen 1800 mg; Test type: Other; p = 0.415, Miettinen & Nurminen; Difference in Percent = -0.9, 95% CI 2-sided [-3.7 to 1.6]
Statistical Analysis 5: Comparison: Etoricoxib 120 mg vs Ibuprofen 1800 mg; Test type: Other; p = 0.965, Miettinen & Nurminen; Difference in Percent = -0.1, 95% CI 2-sided [-3.0 to 2.8]
Statistical Analysis 6: Comparison: Placebo; Placebo vs. Ibuprofen 1800 mg; Test type: Other; p = 0.227, Miettinen & Nurminen; Difference in Percent = 2.3, 95% CI 2-sided [-1.3 to 8.4]
Statistical Analysis 7: Comparison: Etoricoxib 90 mg vs Etoricoxib 120 mg; Test type: Other; p = 0.437, Miettinen & Nurminen; Difference in Percent = 0.8, 95% CI 2-sided [-1.7 to 3.6]

5. Primary Outcome: Percentage of Participants With at Least One Hypertension-Related AE
Description: An AE is defined as any unfavorable and unintended change in the structure, function, or chemistry of the body temporally associated with the use of the study product, whether or not considered related to the use of the product. Any worsening (i.e., any clinically significant adverse change in frequency and/or intensity) of a preexisting condition which is temporally associated with the use of the study product, is also an AE.
Time Frame: Up to 21 days
Population: The analysis population consisted of all randomized patients who received at least one dose of study treatment.
Measure: Number; unit: Percentage of Participants
Arm/Group | Etoricoxib 90 mg | Etoricoxib 120 mg | Ibuprofen 1800 mg | Placebo
Number analyzed (Participants) | 222 | 230 | 223 | 98
Percentage of Participants | 3.6 | 1.3 | 3.1 | 3.1
Statistical Analysis 1: Comparison: Etoricoxib 90 mg vs Placebo; Test type: Other; p = 0.806, Miettinen & Nurminen; Difference in Percent = 0.5, 95% CI 2-sided [-5.3 to 4.5]
Statistical Analysis 2: Comparison: Etoricoxib 120 mg vs Placebo; Test type: Other; p = 0.278, Miettinen & Nurminen; Difference in Percent = -1.8, 95% CI 2-sided [-7.4 to 1.4]
Statistical Analysis 3: Comparison: Ibuprofen 1800 mg vs Placebo; Test type: Other; p = 0.971, Miettinen & Nurminen; Difference in Percent = 0.1, 95% CI 2-sided [-5.7 to 3.9]
Statistical Analysis 4: Comparison: Etoricoxib 90 mg vs Ibuprofen 1800 mg; Test type: Other; p = 0.786, Miettinen & Nurminen; Difference in Percent = 0.5, 95% CI 2-sided [-3.2 to 4.2]
Statistical Analysis 5: Comparison: Etoricoxib 120 mg vs Ibuprofen 1800 mg; Test type: Other; p = 0.184, Miettinen & Nurminen; Difference in Percent = -1.8, 95% CI 2-sided [-5.2 to 1.0]
Statistical Analysis 6: Comparison: Placebo; Placebo vs. Ibuprofen 1800 mg; Test type: Other; p = 0.971, Miettinen & Nurminen; Difference in Percent = -0.1, 95% CI 2-sided [-3.9 to 5.7]
Statistical Analysis 7: Comparison: Etoricoxib 90 mg vs Etoricoxib 120 mg; Test type: Other; p = 0.113, Miettinen & Nurminen; Difference in Percent = -2.3, 95% CI 2-sided [-5.8 to 0.6]

6. Primary Outcome: Percentage of Participants With at Least One Opioid-Related AE
Description: An AE is defined as any unfavorable and unintended change in the structure, function, or chemistry of the body temporally associated with the use of the study product, whether or not considered related to the use of the product. Any worsening (i.e., any clinically significant adverse change in frequency and/or intensity) of a preexisting condition which is temporally associated with the use of the study product, is also an AE. Opioid-related AEs include nausea, vomiting, constipation, somnolence, respiratory depression, urinary retention and ileus.
Time Frame: Up to 21 days
Population: The analysis population consisted of all randomized patients who received at least one dose of study treatment.
Measure: Number; unit: Percentage of Participants
Arm/Group | Etoricoxib 90 mg | Etoricoxib 120 mg | Ibuprofen 1800 mg | Placebo
Number analyzed (Participants) | 222 | 230 | 223 | 98
Percentage of Participants | 34.7 | 36.5 | 36.3 | 41.8
Statistical Analysis 1: Comparison: Etoricoxib 120 mg vs Placebo; Test type: Other; p = 0.365, Miettinen & Nurminen; Difference in Percent = -5.3, 95% CI 2-sided [-17.0 to 6.0]
Statistical Analysis 2: Comparison: Etoricoxib 90 mg vs Placebo; Test type: Other; p = 0.222, Miettinen & Nurminen; Difference in Percent = -7.2, 95% CI [-18.8 to 4.2]
Statistical Analysis 3: Comparison: Ibuprofen 1800 mg vs Placebo; Test type: Other; p = 0.349, Miettinen & Nurminen; Difference in Percent = -5.5, 95% CI 2-sided [-17.2 to 5.9]
Statistical Analysis 4: Comparison: Etoricoxib 120 mg vs Ibuprofen 1800 mg; Test type: Other; p = 0.965, Miettinen & Nurminen; Difference in Percent = 0.2, 95% CI 2-sided [-8.7 to 9.0]
Statistical Analysis 5: Comparison: Etoricoxib 90 mg vs Ibuprofen 1800 mg; Test type: Other; p = 0.718, Miettinen & Nurminen; Difference in Percent = -1.6, 95% CI 2-sided [-10.5 to 7.3]
Statistical Analysis 6: Comparison: Placebo; Placebo vs. Ibuprofen 1800 mg; Test type: Other; p = 0.349, Miettinen & Nurminen; Difference in Percent = 5.5, 95% CI 2-sided [-5.9 to 17.2]
Statistical Analysis 7: Comparison: Etoricoxib 90 mg vs Etoricoxib 120 mg; Test type: Other; p = 0.684, Miettinen & Nurminen; Difference in Percent = 1.8, 95% CI 2-sided [-7.0 to 10.6]

7. Secondary Outcome: Average Change From Baseline for Pain Intensity at Rest Over Days 1 to 3 (Etoricoxib vs. Ibuprofen)
Description: The pain intensity difference was measured at rest over Days 1 through 3 in participants treated with etoricoxib (120 mg, 90 mg) compared to ibuprofen for the treatment of pain following total knee replacement orthopedic surgery. Pain intensity difference at rest was measured on a numerical rating scale (NRS) from 0 - 10 points (0=no pain, to 10=pain as bad as you can imagine). Comparison to ibuprofen was conducted in a step-down manner (the 90-mg dose was evaluated only if the null hypotheses for co-primary endpoints [Pain Intensity Difference (PID) and morphine] 120-mg doses were rejected). The primary analyses for change from baseline in average pain intensity at rest over Days 1 to 3 was performed using the longitudinal data analysis (LDA) method with the terms for baseline pain intensity (moderate or severe), type of anesthesia (spinal or general), treatment, day, and the interaction of day by treatment.
Time Frame: Baseline and Days 1-3
Population: All randomized participants, excluding those who didn't receive at least 1 dose of study treatment, lacked 1 post-randomization measurement, were randomized at a specific site, or received continuous infusion of morphine by patient control analgesia (PCA). Per protocol, the placebo arm was not included in this outcome measure.
Measure: Least Squares Mean (95% Confidence Interval); unit: Score on a scale
Arm/Group | Etoricoxib 90 mg | Etoricoxib 120 mg | Ibuprofen 1800 mg
Number analyzed (Participants) | 211 | 224 | 216
Score on a scale | -3.93 [-4.17 to -3.69] | -3.87 [-4.11 to -3.64] | -3.83 [-4.07 to -3.59]
Statistical Analysis 1: Comparison: Etoricoxib 120 mg vs Ibuprofen 1800 mg; Test type: Non-Inferiority — Non-inferiority reached if the upper bound of the 95% confidence interval of the between-treatment difference (Etoricoxib minus Ibuprofen) in LS means is no greater than 1; Difference in Least Squares Mean = -0.04, 95% CI 2-sided [-0.36 to 0.27]
Statistical Analysis 2: Comparison: Etoricoxib 90 mg vs Ibuprofen 1800 mg; Test type: Non-Inferiority — [test comment as in outcome 7, analysis 1]; Mean Difference (Final Values) = -0.10, 95% CI 2-sided [-0.42 to 0.22]

8. Secondary Outcome: Average Total Daily Dose of Postoperative Morphine Over Days 1 to 3 (Etoricoxib vs. Ibuprofen)
Description: The difference in average total daily dose of morphine used over Days 1 through 3 between participants treated with etoricoxib (120 mg, 90 mg) or ibuprofen 1800 mg (administered as 600 mg three times daily, every 8 hours) in the treatment of pain following total knee replacement orthopedic surgery was assessed. Opioids taken were converted to mg morphine equivalents according to the following conventions:1 mg morphine sulphate = 1 mg morphine, 1 mg morphine hydrochloride = 1.17 mg morphine. A 5 mg oxycodone tablet = 2.5 mg morphine,12.5 mg meperidine = 1.67 mg morphine.
Time Frame: Days 1-3
Population: as for outcome 7
Measure: Geometric Least Squares Mean (95% Confidence Interval); unit: milligrams (mg)
Arm/Group | Etoricoxib 90 mg | Etoricoxib 120 mg | Ibuprofen 1800 mg
Number analyzed (Participants) | 215 | 225 | 217
milligrams (mg) | 8.87 [7.88 to 9.97] | 9.25 [8.26 to 10.4] | 8.82 [7.85 to 9.91]
Statistical Analysis 1: Comparison: Etoricoxib 120 mg vs Ibuprofen 1800 mg; Test type: Other — Estimate from ANOVA model with terms for baseline pain intensity, type of anesthesia, treatment, day, and interaction of day by treatment; Between-Treatment Ratio = 1.05, 95% CI 2-sided [0.89 to 1.23] — A ratio <1 indicates a beneficial effect of Etoricoxib
Statistical Analysis 2: Comparison: Etoricoxib 90 mg vs Ibuprofen 1800 mg; Test type: Other — [test comment as in outcome 8, analysis 1]; Between-Treatment Ratio = 1.01, 95% CI 2-sided [0.85 to 1.18] — A ratio <1 indicates a beneficial effect of Etoricoxib
Statistical Analysis 3: Comparison: Etoricoxib 90 mg vs Etoricoxib 120 mg; Test type: Other — [test comment as in outcome 8, analysis 1]; Between-Treatment Ratio = 1.04, 95% CI 2-sided [0.89 to 1.23] — A ratio <1 indicates a beneficial effect of Etoricoxib

9. Primary Outcome: Percentage of Participants Who Discontinued Study Drug Due to an AE
Description: as for outcome 5
Time Frame: Up to 7 days
Population: The analysis population consisted of all randomized patients who received at least one dose of study treatment.
Measure: Number; unit: Percentage of Participants
Arm/Group | Etoricoxib 90 mg | Etoricoxib 120 mg | Ibuprofen 1800 mg | Placebo
Number analyzed (Participants) | 222 | 230 | 223 | 98
Percentage of Participants | 6.3 | 3.5 | 4.5 | 5.1

ADVERSE EVENTS:
Time Frame: Up to 21 days post surgery
Description: The analysis population consisted of all randomized patients who received at least one dose of study treatment.
Groups:
- Ibuprofen 1800mg: Participants received ibuprofen 600 mg every 8 hours, matching placebo to etoricoxib 120 mg once daily, and matching placebo to etoricoxib 90 mg once daily for 7 days.
Arm/Group | Placebo | Etoricoxib 90 mg | Etoricoxib 120 mg | Ibuprofen 1800mg
All-Cause Mortality (participants affected / at risk) | 0/98 | 0/222 | 0/230 | 0/223
Serious Adverse Events (participants affected / at risk) | 4/98 | 5/222 | 4/230 | 5/223
Other Adverse Events (participants affected / at risk) | 57/98 | 110/222 | 116/230 | 108/223
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=98) | Etoricoxib 90 mg (N=222) | Etoricoxib 120 mg (N=230) | Ibuprofen 1800mg (N=223)
Acute myocardial infarction (Cardiac disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Cardiac arrest (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Sinus tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Constipation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Peptic ulcer haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Bacterial infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Bronchitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cellulitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Urinary tract infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Wound infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Anaemia postoperative (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Transient ischaemic attack (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Renal failure (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=98) | Etoricoxib 90 mg (N=222) | Etoricoxib 120 mg (N=230) | Ibuprofen 1800mg (N=223)
Constipation (Gastrointestinal disorders) | 13 (15) | 26 (27) | 32 (36) | 30 (30)
Dyspepsia (Gastrointestinal disorders) | 8 (9) | 5 (5) | 9 (11) | 10 (11)
Nausea (Gastrointestinal disorders) | 31 (37) | 50 (63) | 56 (78) | 53 (70)
Vomiting (Gastrointestinal disorders) | 13 (15) | 27 (29) | 30 (43) | 33 (37)
Pyrexia (General disorders) | 27 (33) | 13 (13) | 25 (29) | 23 (25)
Dizziness (Nervous system disorders) | 3 (5) | 14 (15) | 15 (23) | 14 (15)
Insomnia (Psychiatric disorders) | 11 (13) | 23 (27) | 21 (26) | 17 (20)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 4 (7) | 14 (15) | 14 (25) | 11 (12)
Pruritus (Skin and subcutaneous tissue disorders) | 4 (4) | 19 (19) | 15 (19) | 17 (17)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The SPONSOR must have the opportunity to review all proposed abstracts, manuscripts, or presentations regarding this study 60 days prior to submission for publication/presentation. Any information identified by the SPONSOR as confidential must be deleted prior to submission. SPONSOR review can be expedited to meet publication guidelines.